CLINICAL TRIAL: NCT00305461
Title: A Pilot Study on the Impact of Two Different Doses of Ciclesonide (160 mcg/Day and 320 mcg/Day) Administered in the Evening on Quality of Life in Patients With Moderate Persistent Asthma.
Brief Title: Effect of Ciclesonide on Quality of Life in Patients With Moderate Persistent Asthma (21 to 65 y) (BY9010/AR-101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/AR-101
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Quality of Life; Ciclesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Ciclesonide 160µg
  Interventions: Drug: Ciclesonide
- 2 (Active Comparator): Ciclesonide 320µg
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide — Effect of Ciclesonide on Quality of Life

SUMMARY:
The aim of the study is to compare the effect of ciclesonide on quality of life, pulmonary function and time to first exacerbation in patients with moderate persistent asthma. Ciclesonide will be administered once daily in the evening at two dose levels. The study duration consists of a baseline period (2 weeks) and a treatment period (8 weeks).

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Good health with the exception of asthma
* Clinical diagnosis of moderate persistent asthma during the last 6 months prior to visit B0
* Pre-treatment with inhaled corticosteroids dose equivalent to 250 - 500 mcg BDP / day at stable dosing during the last 4 weeks prior to visit B0, concomitant or not to short-acting beta2-agonists treatment as rescue medication
* FEV1 ≥ 70% and ≤ 90% predicted measured at least 4 h after the last use of rescue medication at visit B0
* Reversibility ≥ 12% and ≥ 200 mL in B0, B0 or T0, after inhalation of 400 mcg of salbutamol
* Patients compliant to recommended pre-treatment

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Chronic obstructive pulmonary disease (COPD)
* Hospitalization within previous four weeks from baseline
* Hospitalization due to asthma within the last twelve months
* Asthma exacerbation within two months previous to baseline
* History of almost fatal asthma at any moment
* Pregnancy, breast feeding, intention to become pregnant during the course of the study or lack of safe contraception in pre-menopausal women
* Exacerbation of asthma within 2 months prior to entry into the baseline period
* Use of systemic steroids up to 2 months (injectable depot steroids 6 months) before entry into the baseline period, or more than 3 times during the last 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
differences in Quality of Life from AQLQ(S) (T end versus T0) | 8 weeks
time to first exacerbation | 8 weeks
differences in FEV1 and FVC from spirometry (T end vs T0). | 8 weeks

SECONDARY OUTCOMES:
percentage of days on which patients perceived asthma control | 8 weeks
percentage of asthma symptoms free days | 8 weeks
percentage of rescue medication-free days | 8 weeks
percentage of nocturnal awakening-free days | 8 weeks
asthma symptom score (daytime score, nighttime score, total score) | 8 weeks
use of rescue medication | 8 weeks
PEF from spirometry | 8 weeks
morning and evening PEF from diary | 8 weeks
diurnal PEF fluctuation. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (6):
- Argentina (6):
  - Altana Pharma/Nycomed, Buenos Aires
  - Altana Pharma/Nycomed, Cap. Fed.
  - Altana Pharma/Nycomed, Córdoba
  - Altana Pharma/Nycomed, Mendoza
  - Altana Pharma/Nycomed, San Miguel de Tucumán
  - Altana Pharma/Nycomed, Santa Fe

REFERENCES:
- See also: BY9010-AR-101-RDS-2009-06-19.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4506&filename=BY9010-AR-101-RDS-2009-06-19.pdf